CLINICAL TRIAL: NCT07054762
Title: Effects of Omega-3 Supplementation on Exercise Performance, Body Composition and Appetite Status in Female Athletes: A Single-Blind Randomized Controlled Trial
Brief Title: Effects of Omega-3 Supplementation on Exercise Performance, Body Composition, and Appetite Status in Female Athletes
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Betul Uner (Other)
Responsible Party: Sponsor-Investigator, Betul Uner, Lecturer, MSc, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-40160-196
Record Dates: First submitted 2025-06-18; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Volleyball Players
Keywords: omega-3; volleyball; Woman; Single blind

STUDY DESIGN:
Intervention Model Description: This study was conducted with an experimental, single-blind, randomized, and placebo-controlled design to examine the effects of omega-3 fatty acid supplementation on exercise performance, body composition, and appetite status in female volleyball athletes.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 supplement (Experimental): Participants in the experimental group were given four capsules of omega-3 fatty acids with breakfast every day for 8 weeks.
  Interventions: Dietary Supplement: omega-3 supplements in female athletes
- placebo (Placebo Comparator): Participants in the control group were given a placebo containing maltodextrin with breakfast every day for 8 weeks.
  Interventions: Dietary Supplement: Placebo Group

INTERVENTIONS:
Dietary Supplement: omega-3 supplements in female athletes — Participants in the experimental group were given four capsules of omega-3 fatty acids with breakfast every day for 8 weeks. Each capsule contains 150 mg of omega-3 fatty acids and has a ratio of 60% EPA and 40% DHA. At the beginning of the study, 24-hour food consumption records were taken 8 times, once a week and at the end. In addition, anthropometric measurements, simplified food appetite questionnaire, muscle pain assessment and muscle endurance test were performed at the beginning and end of the study.
  Arms: Omega-3 supplement
Dietary Supplement: Placebo Group — Participants in the control group were given a placebo containing maltodextrin with breakfast every day for 8 weeks. Each capsule contains 250 mg maltodextrin. At the beginning of the study, 24-hour food consumption records were taken 8 times, once a week and at the end of the study. Additionally, anthropometric measurements, a simplified food appetite questionnaire, muscle pain assessment and muscle endurance test were performed at the beginning and end of the study.
  Arms: placebo

SUMMARY:
Volleyball is a sport that requires high performance and aims to increase endurance. The intense training and competition tempo of athletes directs them to special nutritional needs. Omega-3 fatty acids, in particular, are known for their anti-inflammatory properties and positive effects on the cardiovascular system, and provide potential contributions such as supporting exercise performance, reducing stress levels and improving body composition in athletes. However, studies examining the effects of omega-3 on female volleyball players are rare in the literature.

The purpose of this study is to determine the effect of omega-3 supplementation on exercise performance, body composition and appetite status in 2nd league women's volleyball team athletes. The research group consists of female volleyball players over the age of 18. The potential effects of the recommended level of omega-3 supplementation added to the daily nutrition programs of female athletes without changing their routine nutrition programs will be evaluated in the study.

A single-blind placebo method will be used in this experimental and randomized controlled study. After the participants have a diet low in omega-3 for 2 weeks, they will be divided into two groups; The experimental group will be given 2 capsules of omega-3 supplements with breakfast for eight weeks, while the control group will be given a placebo capsule. This study aims to contribute to the literature on the effects of omega-3 supplements on athlete performance and to better understand the role of nutritional supplements on physiological parameters in female volleyball players.

Anthropometric measurements of the athletes will be taken at the beginning of the intervention, every two weeks during the intervention, and at the end of the intervention, and a 24-hour retrospective food consumption record, a simplified nutritional appetite questionnaire, muscle pain assessment, and a muscle endurance test will be applied.

The collected study data will be analyzed using SPSS 20.0 statistical analysis software. The Kolmogorov-Smirnov test will be used to assess the normality of the data. Percentage, mean, and standard deviation calculations will be used in the analysis of the findings obtained in the study; appropriate statistical analyzes will be performed to examine the relationship between the independent variables of the control and experimental groups and exercise performance, body composition, and appetite status.

DETAILED DESCRIPTION:
An athlete is defined as an individual, whether amateur or professional, who receives regular exercise training and participates in official sports competitions, whether young or adult (1). Volleyball is a complex team sport with an average match duration of 60-90 minutes, which imposes different physical and cognitive demands (2). Volleyball is a sport that requires explosive power, endurance and speed. Volleyball athletes use their physical capacities, such as jumping, quick changes of direction and focus, to the maximum. Research shows that volleyball players train three to five days a week and participate in special exercises to increase their muscular endurance and conditioning (3). Volleyball, an open skill sport, requires motor movements characterized by effective visual search and action anticipation in dynamic and complex environments (4). Increased ability for action anticipation is closely associated with the ability to effectively "read the game" and having superior game intelligence (5), which is a prerequisite for successfully applying techniques and tactics (4). Consequently, physical performance, including vertical jump, short-distance agility, and spiking, as well as perceptual-cognitive performance, are key determinants of volleyball performance (6). Fatigue is common in sports, especially in high-intensity, long-duration activities such as volleyball (7). A comprehensive understanding of how fatigue affects action anticipation and physical performance is crucial to developing effective training strategies for top-level volleyball players (8).

Female athletes may have different hormonal structures, training responses, and muscle recovery processes. In this context, it is thought that muscle recovery is slower in female athletes and that they may face a higher risk of inflammation. It is stated that the anterior cruciate ligament injury rates are four to eight times higher in women than in men (9). It is thought that female volleyball players need additional support to prevent muscle damage during their weekly training and match periods, especially during intense training periods (8).

Omega-3 polyunsaturated fatty acids (PUFA) cannot be produced by the human body, so it is important to get them through diet or supplements. There are three main omega-3 fatty acids: alpha-linolenic acid (ALA, 18:3 n-3), eicosapentaenoic acid (EPA, 20:5 n-3), and docosahexaenoic acid (DHA, 22:6 n-3). ALA is found in plant-based sources such as flaxseed, chia seeds, and walnuts, while EPA and DHA are primarily found in seafood and fatty fish such as salmon, tuna, and mackerel (10). The benefits of omega-3 fatty acids are wide-ranging. Omega-3s are thought to have anti-inflammatory and anti-thrombotic properties, lower plasma triglycerides and low-density lipoprotein cholesterol, improve vasomotor and endothelial function, and inhibit cell growth factors (11). Studies have confirmed that omega-3 supplements strengthen memory, reduce symptoms of depression, prevent age-related cognitive decline, and are effective in treating depression (10,12,13).

In athletes, omega-3 fatty acids are particularly notable for their properties such as accelerating muscle repair and recovery, reducing post-exercise inflammation, and increasing endurance. Recently, it has been accepted that omega-3 may play a role in these processes, not only counteracting exercise-induced inflammation but also improving muscle health and energy utilization, and may be used as an ergogenic supplement. It has been shown that it can contribute to a faster recovery process in athletes by reducing post-exercise inflammation and muscle damage, and that it can have positive effects on endurance athletes by increasing muscle protein synthesis in athletes (14). It has been shown that regular omega-3 intake in athletes reduces inflammation levels, supports cardiovascular health, and has positive effects on general health (15). A randomized controlled trial has shown that omega-3 reduces exercise-induced muscle damage in athletes (16).

A review has shown that omega-3 use in team athletes has positive effects on athlete performance (17). Meta-analysis studies have reported that omega-3 use in endurance athletes reduces inflammation and muscle damage markers (18) and muscle pain after exercise (19). It has been stated that omega-3 supplements applied to athletes of both genders are beneficial for skeletal muscle adaptations and body recomposition (20). It has been concluded that omega-3 supplements applied to professional rugby athletes help reduce muscle pain and better preserve explosive power (21). It has been stated that omega-3 fatty acid supplements given to male athletes do not have a significant effect on improving muscle damage (22). It has been reported that omega-3 enriched chicken egg supplements to male athletes reduce oxidative stress and have positive effects against physical stress (23). Studies on female athletes are quite limited in the scientific literature. A randomized controlled study conducted with female athletes has indicated that omega-3 supplements may be effective in the recovery process after training (24).

The effects of omega-3 intake on body composition are still unclear, but they appear to increase muscle synthesis (25, 26) or limit muscle loss (27). A randomized controlled trial has shown that omega-3 supplementation in athletes has positive effects on muscle gain and fat loss (28). In addition, there is no clear standard in the literature regarding EPA and DHA ratios. While most studies have preferred 60% EPA and 40% DHA ratios, some studies have changed these ratios according to the physiological needs of athletes. In particular, it is known that high EPA ratios support inflammation-reducing effects, while DHA has neurological benefits. However, most studies conducted on female athletes have not examined the effects of these proportional differences (29). This is considered an important deficiency in the literature.

This planned study aims to determine the effects of omega-3 supplementation on exercise performance, body composition and appetite status in female volleyball players with a single-blind, randomized and placebo-controlled design.

Hypotheses:

H0a: Given omega-3 supplementation has no effect on exercise performance in women's volleyball team athletes.

H1a: Given omega-3 supplementation has an effect on exercise performance in women's volleyball team athletes.

H0b: Given omega-3 supplementation has no effect on body composition in women's volleyball team athletes.

H1b: Given omega-3 supplementation has an effect on body composition in women's volleyball team athletes.

H0c: Given omega-3 supplementation has no effect on appetite in women's volleyball team athletes.

H1c: Given omega-3 supplementation has an effect on appetite in women's volleyball team athletes.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Participants should not have a chronic disease or regular medication use
* Not have used omega-3 or similar fatty acid supplements in the last 6 months

Exclusion Criteria:

* Having a diet model that is applied regularly
* Having undergone any surgical intervention
* Being in pregnancy or lactation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of omega-3 supplementation given to female volleyball players for 8 weeks on exercise performance. | It lasted 8 weeks. January 10, 2025 - March 17, 2025
  Muscle soreness assessment and muscle endurance test will be performed for exercise performance. Muscle Soreness Assessment is represented by a scale between 0 (no pain) and 10 (extreme pain) while athletes squat against a wall at a 90° angle with their thighs parallel to the ground. Athletes will make a number according to the pain they feel.
  * 0: No Pain
  * 1-3: Mild pain
  * 4-6: Moderate pain
  * 7-9: Severe pain
  * 10: Worst pain Muscle Endurance Test; In order to evaluate the endurance of the abdominal muscles, the maximum number of sit-up repetitions of the participant in one minute is determined and the number of repetitions made during this period indicates the endurance level of the abdominal muscles.
Evaluation of the effects of omega-3 supplementation given to female volleyball players for 8 weeks on body composition. | It lasted 8 weeks. January 10, 2025 - March 17, 2025
  Height, weight, neck, waist, hip circumference measurements will be used to determine body composition. Weight in kilograms and height in meters will be used to calculate BMI. It will be determined whether the applied omega-3 supplement creates any change in the athletes' BMI and fat value (thanks to circumference measurements).
Evaluation of the effect of omega-3 supplementation on appetite status in female volleyball players given for 8 weeks. | It lasted 8 weeks. January 10, 2025 - March 17, 2025
  The athletes' appetite status was assessed using the Simplified Nutrition Appetite Questionnaire. The Simplified Nutrition Appetite Questionnaire consists of four questions. Each question is given a value between one and five points according to its answer. The total score is calculated by adding the points corresponding to the participants' answers, and an increase in the score indicates an increased appetite.

CONTACTS AND LOCATIONS:
Locations (1):
- Muğla Sıtkı Koçman University/Muğla Training and Research Hospital Neurology Polyclinic, Muğla, Mentese, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR